CLINICAL TRIAL: NCT02018107
Title: PET/CT-Guided Liver Tumor Ablation: Intraprocedural Assessment of Results Using Ammonia Perfusion PET
Brief Title: PET/CT-Assessment of Liver Tumor Ablation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Paul Shyn, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 13-464
Record Dates: First submitted 2013-12-17; First posted 2013-12-23 (Estimated); Results first posted 2020-03-26 (Actual); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Liver Tumor; Liver Neoplasms
Keywords: Liver Tumor Ablation; Liver Neoplasms; Positron Emission Tomography; Computed Tomography
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms | interventions — Positron-Emission Tomography

STUDY DESIGN:
Intervention Model Description: This is a diagnostic imaging study, involving FDA-approved radiopharmaceuticals. Applying a "Phase" to the study is N/A, even though the Study Phase had to be entered above.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- N-13 ammonia to image liver PET perfusion (Experimental): This single-arm study involves the non-therapeutic administration of a radiopharmaceutical, N-13 ammonia or F-18 fluorodeoxyglucose, one to two doses, during the tumor ablation procedure. The N-13 ammonia perfusion PET scan is a diagnostic imaging test. The tumor ablation procedure is performed according to our standard clinical practice and is not itself a research activity. The use of N-13 ammonia to image liver perfusion with a PET scanner is the research portion of the procedure. The participant will receive one or two IV doses of N-13 ammonia (10 mCi/dose) for intraprocedural assessment of ablation results. Not more than two doses will be administered and one or both doses will be administered on the day of the tumor ablation procedure only
  Interventions: Diagnostic Test: N-13 ammonia or F-18 fluorodeoxyglucose; Diagnostic Test: PET scan

INTERVENTIONS:
Diagnostic Test: N-13 ammonia or F-18 fluorodeoxyglucose — PET tracer
Diagnostic Test: PET scan — PET scan

SUMMARY:
In this research study, the investigators are evaluating whether ammonia PET scans or FDG PET perfusion scans are more useful in helping radiologists determine whether liver tumors were successfully destroyed by the heating or freezing procedures (ablations) than other scans currently available to radiologists, such as CT scans and MRI scans.

The currently available scan (usually a CT scan with contrast dye) is not always effective in showing how completely the tumor has been destroyed. The ammonia PET scan is a different way of looking at how much tumor has been destroyed. This study will compare the standard scan (CT scan) with the ammonia PET scan.

DETAILED DESCRIPTION:
The plan for this study involves the non-therapeutic administration of a radiopharmaceutical, N-13 ammonia or F-18 fluorodeoxyglucose, one to two doses, during the tumor ablation procedure. The perfusion PET scan is a diagnostic imaging test. The tumor ablation procedure is performed according to our standard clinical practice and is not itself a research activity. The use of N-13 ammonia or F-18 fluorodeoxyglucose to image liver perfusion with a PET scanner is the research portion of the procedure. The patient will receive one or two doses of N-13 ammonia (10 mCi (millicurie)/dose) for intraprocedural assessment of ablation results. Not more than two doses will be administered and one or both doses will be administered on the day of the tumor ablation procedure only. The ammonia perfusion scan will not be used to change or modify the ablation procedure.

After the screening procedures confirm that that the participant is eligible to participate in the research study:

* Ammonia Perfusion PET: The participant will be scheduled for the tumor ablation procedure as part of the participant's routine care. If the participant decided to take part in this research study, then the participant will have one or two ammonia perfusion PET scans during the ablation procedure to see if the ablation was successful or not as compared to standard CT scanning. The ammonia perfusion PET scans are the research part of the participant's procedure. The rest of the participant's procedure is not research. The participant will receive one or two doses of the radioactive tracer called N-13 ammonia. This tracer is administered through the same IV (thin tube placed in a vein) used by the Anesthesiologist to give the participant routine medications that relax the participant, prevent pain, and allow the participant to sleep during the procedure. This tracer does not treat the participant's tumor in any way. Instead, the tracer may allow the radiologist to better see how much of the participant's tumor was destroyed.
* Photographs: Photographs may be taken during the procedure. Care will be taken to ensure these do not reveal the participant's identity.
* Clinic visits: The investigators routinely see patients after tumor ablation procedures within one to two weeks after the procedure and then every three months after the procedure for one to two years, and as needed in the future. Accordingly, the clinic visits are routine and not an added research commitment.

ELIGIBILITY:
Inclusion Criteria:

* Adults, 18 years or older
* Referral from an internist, oncologist, or surgeon for liver tumor ablation consultation
* ECOG (Eastern Cooperative Oncology Group) Performance Status < 3
* Liver tumor ablation judged to be appropriate based on clinical assessment in the BWH (Brigham & Women's Hospital) Tumor Ablation Clinic by the tumor ablation interventional radiologist, per standard clinical practice
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Uncorrectable coagulopathy (due to bleeding risk)
* Pulmonary disease precluding monitored anesthesia care or general anesthesia
* Severe renal insufficiency, EGFR (estimated glomerular filtration rate) < 30
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, significant cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Childs-Pugh Class C cirrhosis
* Occlusive main portal vein thrombosis
* Presence of biliary-enteric anastomosis (due to risk of biliary infection)
* Pregnant women are excluded (because both CT and PET/CT scans involve the use of ionizing radiation which may pose a potential teratogenic effect on the fetus.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2014-01; Primary Completion 2018-02-16 (Actual); Study Completion 2019-02-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul B. Shyn, M.D., Principal Investigator — Brigham and Women's Hospital
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

REFERENCES:
- [Derived] Shyn PB, Cubre AJ, Catalano PJ, Lee LK, Hyun H, Tuncali K, Seol JG, Levesque VM, Gerbaudo VH, Kapur T, Chao RT, Silverman SG. F-18 FDG perfusion PET: intraprocedural assessment of the liver tumor ablation margin. Abdom Radiol (NY). 2021 Jul;46(7):3437-3447. doi: 10.1007/s00261-021-02970-8. Epub 2021 Feb 19. PMID 33606061

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 33 unique participants were enrolled and consented for this study, 6 participants were then excluded from the study.
  Thus, the count of subjects is 27 who were assigned to intervention. Out of 27 participants, 1 subject participated in both interventions.
Pre-assignment Details: 33 unique participants were enrolled and consented for this study, 6 participants were then excluded from the study.
  Thus, the count of subjects is 27. Out of 27 participants, 1 subject participated in both interventions.
Period: Overall Study
Arm/Group | N-13 Ammonia to Image Liver PET Perfusion
Started | 27
Completed | 27
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: There were 27 unique participants and one participant participated twice (in both interventions).
Groups:
- N-13 Ammoniaor F-18 Fluorodeoxygl to Image Liver PET Perfusion: This single-arm study involves the non-therapeutic administration of a radiopharmaceutical, N-13 ammonia or F-18 fluorodeoxyglucose, one to two doses, during the tumor ablation procedure. The N-13 ammonia perfusion PET scan is a diagnostic imaging test. The tumor ablation procedure is performed according to our standard clinical practice and is not itself a research activity. The use of N-13 ammonia to image liver perfusion with a PET scanner is the research portion of the procedure. The participant will receive one or two IV doses of N-13 ammonia (10 mCi/dose) for intraprocedural assessment of ablation results. Not more than two doses will be administered and one or both doses will be administered on the day of the tumor ablation procedure only
  N-13 ammonia or F-18 fluorodeoxyglucose: PET tracer
  PET scan: PET scan
Arm/Group | N-13 Ammoniaor F-18 Fluorodeoxygl to Image Liver PET Perfusion
Number analyzed (Participants) | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 14
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 27

OUTCOME MEASURES:

1. Primary Outcome: Number and Percentage of Tumors With Complete, Circumferential Ablation Margin Visibility During FDG PET/CT-guided Liver Ablations (AP-PET-1 v. Contrast-enhanced MRI)
Description: For FDG-avid tumors, compare the rates of complete, circumferential ablation margin visibility during FDG PET/CT-guided liver ablations using two imaging techniques: intra-procedural AP-PET-1(research scan #1) and post-procedural contrast enhanced MRI . Discordance rates for complete ablation margin visibility between the two imaging techniques will be calculated.
Time Frame: 2 Years
Population: In this study, the number of tumors were analysed. There 8 participants with 11 tumors that were analysed for N-13 ammonia to image liver PET perfusion and 31 tumors in 20 patients were analysed in F-18 fluorodeoxyglucose to image liver PET perfusion. 1 participant participated in both interventions. Total unique participants 27.
Measure: Count of Units; unit: Tumors
Units Other Than Participants: Tumors
Groups:
- N-13 Ammonia or F-18 to Image Liver PET Perfusion: This single-arm study involves the non-therapeutic administration of a radiopharmaceutical, N-13 ammonia or F-18 fluorodeoxyglucose, one to two doses, during the tumor ablation procedure. The N-13 ammonia perfusion PET scan is a diagnostic imaging test. The tumor ablation procedure is performed according to our standard clinical practice and is not itself a research activity. The use of N-13 ammonia to image liver perfusion with a PET scanner is the research portion of the procedure. The participant will receive one or two IV doses of N-13 ammonia (10 mCi/dose) for intraprocedural assessment of ablation results. Not more than two doses will be administered and one or both doses will be administered on the day of the tumor ablation procedure only
  N-13 ammonia or F-18 fluorodeoxyglucose: PET tracer
  PET scan: PET scan
Arm/Group | N-13 Ammonia or F-18 to Image Liver PET Perfusion
Number analyzed (Participants) | 27
Number analyzed (Tumors) | 42
Tumors
  Total Tumors | 42
  Assessibility of ablation margin by Pet Perfusion | 40
  Assessibility of ablation margin by MRI | 25

2. Secondary Outcome: Does an Inadequate Ablation Margin on PET Predict Local Progression? Compare to MRI?
Description: Percentage of tumors with an inadequate margin on PET that progressed locally? Compare to MRI?
Time Frame: 2 Years
Measure: Number; unit: percentage of tumors
Units Other Than Participants: Tumors
Arm/Group | N-13 Ammonia or F-18 to Image Liver PET Perfusion
Number analyzed (Participants) | 27
Number analyzed (Tumors) | 42
percentage of tumors
  PET:% local progression based on inadequate margin | 53.84
  MRI:% local progression based on Inadequate margin | 83.33
  PET: % local non-progression per adequate margin | 96.29
  MRI: % local non-progression per adequate margin | 89.47

ADVERSE EVENTS:
Time Frame: 3 months
Description: 27 participants were at risk
Arm/Group | N-13 Ammonia to Image Liver PET Perfusion
All-Cause Mortality (participants affected / at risk) | 0/27
Serious Adverse Events (participants affected / at risk) | 0/27
Other Adverse Events (participants affected / at risk) | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-01): https://cdn.clinicaltrials.gov/large-docs/07/NCT02018107/Prot_SAP_000.pdf